CLINICAL TRIAL: NCT04335240
Title: Premature Family Music Therapy Intervention (PFMI): an Italian Protocol to Support Parenting, Attachment Bond and Preterm Development
Brief Title: Premature Family Music Therapy Intervention (PFMI)
Acronym: PFMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Barbara Sgobbi, Principal Investigator, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Music Therapy
Keywords: Music therapy; NICU; Preterm; Infants; Music; HRV; Neurodevelopment
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: A prospective randomized controlled trial will be conducted. Infants will be divided in two subgroups: an intervention group (that will undergo music therapy treatment) and a control group. To evaluate the effectiveness of the protocol, the effects of treatment in the short- and long-term period will be evaluated, with particular reference to the clinical course, the neuro-behavioral development of the premature baby and the relationship with his parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Intervention (Experimental): This protocol is a Family Centered Care Music Therapy Intervention. The methodologies will provide early intervention from the first days of hospitalization in NICU and consist of music therapy sessions both "active" (parental chant, live music and lullaby) and "receptive" (listening to recorded tracks). The music therapy accompanies the newborn and the parents during the hospitalization and focuses its attention on the emotional-relational care, according to the different needs that they will develop over time.Therapy sessions will be performed starting from three times per week, on three different days of the week, during the entire hospitalization of the enrolled infants. After discharge music therapy treatment will be performed once a week until twelve months of corrected age.
  Stress level of infants and parents and neurobehavioral and neurological development of children will be assessed.
  Interventions: Other: Premature family music therapy intervention to support parenting, attachment bond and preterm development
- No music therapy intervention (No Intervention): Music therapy is not administered in this group. Control group (no music therapy). During the entire hospital stay, newborn babies will receive standard care in use in the neonatal intensive care unit.

INTERVENTIONS:
Other: Premature family music therapy intervention to support parenting, attachment bond and preterm development — We have structured an integrated psychological and music therapeutic protocol that aims to limit or overcome neonatal long-term developmental morbidities, promote parenting and attachment bond in preterm infants.
  Arms: Music Therapy Intervention

SUMMARY:
The music therapy intervention it is dedicated to premature baby and their family at the Neonatal Intensive Care Unit (NICU)of the Woman-Child department "Hospital Del Ponte". In NICU an integrated psychological and music therapeutic protocol has been structured. The protocol aims to limit or overcome long-term developmental morbidities, promote parenting and attachment bond in preterm infants. Protocol is named "Premature family music therapy intervention (PFMI): an Italian protocol to support parenting, attachment bond and preterm development". The methodologies will provide early intervention from the first days of hospitalization in NICU and use music therapy sessions "active" (chant parental, live music and lullaby) and "receptive" (listening to recorded tracks). Such therapy becomes a support for the born prematurely and her parents during hospitalization and after discharge. The music therapy accompanies the newborn and his parents during the hospitalization and focuses its attention on the emotional-relational care, according to the different needs of babies and parents.

This protocol it is a Family Centered Care Music Therapy Intervention.

DETAILED DESCRIPTION:
All infants will be enrolled when in stable clinical condition within two weeks after birth. Therapy sessions will take place minimum three times per week on three different days of the week directly at the unit during the entire hospitalization until discharge. After discharge music therapy treatment will be performed once a week until twelve months of corrected age.

The infant's wellbeing and relaxation during each session of music therapy will be measured using the following parameters:

HRV (Heart Rate Variability) analysis Oxygen's saturation Stress level of the child

Infants will be followed till 12 months of corrected age. Investigators will assess:

Neuro-behavioral and neurological development of the child Stress level of the parents

ELIGIBILITY:
Inclusion Criteria, Preterm infants born, will be eligible for the study, if they will be:

1. Born between 22+6- and 32-weeks postmenstrual age
2. Weight less than 1500 g
3. Free from major congenital defects
4. Free from cerebral and/or intraventricular hemorrhage
5. Singleton or twin gestation
6. No sensorineural hearing loss (at discharge, passed bilateral hearing screening)
7. Free from Necrotizing enterocolitis
8. Free from severe retinopathy
9. No asphyxiated

11. No terms of surgical relevance 12. Born from HIV negative and drug free mothers

Exclusion Criteria, we will exclude infants whose mothers will be:

1. Affected by drug dependence
2. Affected by psychosis or other severe mental health problems
3. Unable to adequately speak/understand Italian language
4. Younger than 18 years of age
5. Physically unable to participate

Ages: 23 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
HRV analysis | through test completion, starting from 5 minutes before the test until 5 minutes after test ended
  The heart rate variability is related to the interaction of the sympathetic nervous system (alarm system) and parasympathetic (vagal). HRV derives from the balance of Low Frequency (LF) and High Frequency (HF). LF parameter represents the Sympathetic System and is correlated to a state of stress, while HF parameter represents the Parasympathetic System and is correlated to a state of relaxation. The balance of the two parameters (represented by value 1), means that their relationship is a state of well-being.
Oxygen's saturation | through test completion, starting from 5 minutes before the test until 5 minutes after test ended
  Monitor oxygen saturation by medical monitor in Neonatal Intensive Care and Neonatology.

SECONDARY OUTCOMES:
Stress level of the parents | at 6 and 12 months of corrected age
  Parenting Stress Index-Short Form (PSI-SF, Abidin, 1995; Italian version edited by Guarino et al., 2007) at 6-12 months of corrected age State-Trait Anxiety Scale (STAI; Spielberger, 1983; Italian validation of Pedrabissi and Santinello (1996) at 6-12 months of corrected age Beck Depression Inventory (BDI, Beck, 1967) at 6-12 months of corrected age
Neuro-behavioral and neurological development of the child | at 6-12 months of corrected age
  Temperament detected by the test QUIT (Italian Questionnaires of Temperament Axia, 2002)
Neuro-behavioral and neurological development of the child | at 1-3-6-9-12 months of corrected age.
  General movements (GM). Using digital recording and analysis.
Neuro-behavioral and neurological development of the child | 12 months of corrected age
  Griffiths Scale

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Agosti, MD, Principal Investigator — Neonatologia, TIN e Pediatria Verbano- Ospedale F. del Ponte
Locations (1):
- Ospedale F. Del Ponte, Varese, Italy

IPD SHARING:
Plan to Share IPD: No